CLINICAL TRIAL: NCT04049877
Title: Retrospective and Prospective Disease Progression and Quality of Life in X-linked Hypophosphatemia (XLH)
Brief Title: Retrospective and Prospective Disease Progression and Quality of Life in XLH
Status: Completed | Type: Observational
Sponsor: Medialis Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: Med_Asst19
Record Dates: First submitted 2019-08-07; First posted 2019-08-08 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: X-linked Hypophosphatemia (XLH)
MeSH Terms: conditions — Familial Hypophosphatemic Rickets

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: None - Observational study — None - Observational study

SUMMARY:
There is limited empirical data documenting disease progression and impact on quality of life for patients with X-linked hypophosphatemia (XLH). This study seeks to investigate the impact of XLH in adults living in the UK retrospectively and prospectively over a 12 month period, using qualitative interviews, SEIQoL-DW, EQ-5D-5L, SF36 quality of life tools.

XLH is a rare, genetic, chronically debilitating and deforming condition (www.nice.org.uk/guidance/HST8). XLH is characterised by renal phosphate wasting, hypophosphatemia and defective bone mineralisation. The incidence of XLH is reported to be between 1:20,000 and 1:25,000 live births. In the UK, it is estimated that there are around 250 paediatric XLH patients and around 2,500 adult XLH patients (Delmestri,et al [Unpublished report]2018). The clinical phenotype of XLH is varied amongst patients, even among affected members of the same family. This can range from no signs or symptoms, slow growth in children, short stature, bone abnormalities that can affect movement and result in pain, bowed legs and knocked knees (where lower legs are positioned at an outward angle), tooth abscesses and excessive dental caries and hearing loss (adult patients only).

This study will recruit 36 adults living with XLH, who are aged 28 years or over and living in the UK. The study will be advertised by the Sponsor and funder Medialis Ltd and via the patient organisation Metabolic Support UK. All study activities will take place via tele-visits and online questionnaires. The study will last approximately 2 years, allowing for one-year recruitment and a further 12 months to conduct all study visits.

ELIGIBILITY:
Inclusion Criteria:

* • Participant has a diagnosis of XLH

  * Participant is aged 28 years and above.
  * Participant is capable of providing informed consent
  * Participant is able to read and converse in English
  * Participant is able to comply with the study schedule (5 tele-visits over a 12-month period)

Exclusion Criteria:

* • Participant does not have a diagnosis of XLH

  * Participant is aged under 28 years
  * Participant is not capable of giving informed consent
  * Participant is unable to read and converse in English
  * Participant is unable to comply the with study schedule (5 tele-visits over a 12-month period)

Min Age: 28 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults with XLH
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2019-07-07 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-07-28 (Actual)

PRIMARY OUTCOMES:
Schedule for the Evaluation of Individual Quality of Life Direct Weight (SEIQoL-DW) | 12 months
  Change in quality of life
Disease progression in adults living with XLH | 12 months
  Qualitative investigation of disease progression

SECONDARY OUTCOMES:
EQ- 5D-5L | 12 months
  Quality of life measure
SF36 | 12 months
  Quality of life measure

CONTACTS AND LOCATIONS:
Locations (1):
- Medialis, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: This is a link to the publication resulting from this study. — https://ojrd.biomedcentral.com/articles/10.1186/s13023-020-01434-4